CLINICAL TRIAL: NCT01834170
Title: EUS-guided Intratumoral Gemcitabine Therapy in Locally Advanced Unresectable Pancreatic Cancer: A Phase 1 Study
Brief Title: EUS-guided Intratumoral Gemcitabine in Locally Advanced Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Tehran (Other)
Responsible Party: Principal Investigator, Mehdi Mohamadnejad, Assistant Professor of Medicine, University of Tehran
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DDRC 92-1
Record Dates: First submitted 2013-04-06; First posted 2013-04-17 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic cancer; Pancreatic adenocarcinoma; Endoscopic ultrasound
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intratumoral gemcitabine injection (Experimental): Intratumoral injection of gemcitabine by means of endoscopic ultrasound.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — Two intratumoral injections of gemcitabine under endoscopic ultrasound (EUS)-guidance at month 0 and month 3.
  The patients will receive systemic chemotherapy with or without radiotherapy at the discretion of oncologist
  Other Names: Gemzar

SUMMARY:
Pancreatic cancer is the 11th most common type of cancer but it is the fourth leading cause of cancer death. The only effective treatment for pancreatic cancer includes surgery. However, only 20% of the patients have surgically treatable disease. Also, the 5-year survival for the surgically treated patients is only 15%.

About 40% of the patients present with advanced disease with distant metastasis, and the remaining 40% present with locally advanced unresectable cancer with the tumor invaded into surrounding major vessels. For those with locally advanced disease, systemic chemotherapy with or without radiotherapy provides palliation of the symptoms but cannot cure the disorder. Systemic chemotherapy is given through peripheral vessels.

The investigators hypothesized that direct injection of the chemotherapeutic drug into the tumor may help to boost the effect of systemic chemotherapy and radiotherapy in those with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
In this study, gemcitabine will be injected directly into the tumor by means of endoscopic ultrasound (EUS) in the eligible patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically verified pancreatic adenocarcinoma who have locally advanced unresectable tumor

Exclusion Criteria:

* Early stage resectable pancreatic cancer with the intact surrounding major vessels on imaging
* Pancreatic cancer with distant metastasis
* Unwilling to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 6 months

SECONDARY OUTCOMES:
Proportion of participants who remain alive one year after enrollment compared to the historical matched control group | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Mohamadnejad, M.D., Principal Investigator — Digestive Disease Research Center, University of Tehran/Medical sciences; Reza Malekzadeh, M.D., Study Chair — Digestive Disease Research Center, University of Tehran/Medical Sciences
Locations (1):
- Digestive Disease Research Center, Shariati ospital, Tehran, Iran